CLINICAL TRIAL: NCT03903666
Title: Anomalies of Nocturnal Gaz Exchanges in Patients With Down Syndrome Aged From 4 to 16 Years
Brief Title: Anomalies of Nocturnal Gaz Exchanges in Patients With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Jerome Lejeune (Other)
Collaborators: Hôpital Armand Trousseau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TriRespi
Record Dates: First submitted 2019-03-23; First posted 2019-04-04 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Down Syndrome
Keywords: Sleep Apnoa; Down Syndrome; Children; OSA
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Down syndrome patients aged from 4 to 16 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Experimental): 47 Down syndrome patients age from 4 to 16
  Interventions: Other: Nocturnal gaz exchanges measurement

INTERVENTIONS:
Other: Nocturnal gaz exchanges measurement — Nocturnal gaz exchanges at patient's home BRIEF neuropsychological questionnaire VINELAND-II neuropsychological questionnaire Clinical OSA assessment Dysautonomia assessment

SUMMARY:
Recently, retrospective studies have shown that Down Syndrome children have a higher CO2 (carbone dioxide) sleep pressure than the general pediatric population. This increase does not seem to be always related to sleep apnea. The Investigators wish to confirm these results prospectively. The investigators hypothesize that this alveolar hypoventilation may be due to ventilatory control disorders caused by dysautonomia, but also to a decrease in the strength of the respiratory muscles within the framework of the global muscular hypotonia described in children with Down syndrome. .

DETAILED DESCRIPTION:
47 Down syndrome patients age from 4 to 16 will be included. They will perform a medical visit at J0, then a measurement of gaz nocturnal exchanges at home within 1 month

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome patient without mosaicism
* Age 4 to 16 years
* Predominant French language in the living environment

Exclusion Criteria:

* OAS diagnostic focused on an earlier polysomnography
* Methylphenidate treatment started before inclusion

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with high mean PtcCO2 as assessed by nocturnal gas exchange recordings | 2 months

SECONDARY OUTCOMES:
Percentage of total sleep time with a PtcCO2 in mmHg higher than 50; mean, maximum and minimum SpO2 in % | 2 months
Number of patients with low mean, minimum and maximum SpO2 (oyxygen saturation) and/or % of Total sleep time spent with a PtcCO2 higher than 50 mmHg, higher than 20%, as measured by nocturnal gas exchange recordings. | 2 months
Correlation between nocturnal PtcCO2 value and the existence of executive function and behavioral disorders assed by the Dysautonomia questionnaire | 2 months
Correlation between nocturnal PtcCO2 value and the existence of executive function and behavioral disorders measured by Hand Grip assessment | 2 months
Correlation between nocturnal PtcCO2 value and the existence of executive function and behavioral disorders measured by OSA (Obstructive Sleep Apnea) assessment questionnaire | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: TAYTARD MD Jessica, Principal Investigator — Hôpital Armand Trousseau
Locations (1):
- Hôpital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman JL, Del Negro CA, Gray PA. Understanding the rhythm of breathing: so near, yet so far. Annu Rev Physiol. 2013;75:423-52. doi: 10.1146/annurev-physiol-040510-130049. Epub 2012 Oct 29. PMID 23121137
- [Background] Trang H, Brunet JF, Rohrer H, Gallego J, Amiel J, Bachetti T, Fischbeck KH, Similowski T, Straus C, Ceccherini I, Weese-Mayer DE, Frerick M, Bieganowska K, Middleton L, Morandi F, Ottonello G; European Central Hypoventilation Syndrome Consortium. Proceedings of the fourth international conference on central hypoventilation. Orphanet J Rare Dis. 2014 Dec 5;9:194. doi: 10.1186/s13023-014-0194-5. PMID 25928806
- [Background] Ng DK, Hui HN, Chan CH, Kwok KL, Chow PY, Cheung JM, Leung SY. Obstructive sleep apnoea in children with Down syndrome. Singapore Med J. 2006 Sep;47(9):774-9. PMID 16924359